CLINICAL TRIAL: NCT00167128
Title: The Phonak EduLink-System in Students With Specific Performance Deficits in Speech-in-Noise Intelligibility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Phonak AG, Switzerland (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: phonpaed002
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2007-08-15 (Estimated); Status verified 2006-05

CONDITIONS: Auditory Processing Disorder
Keywords: Auditory Processing Disorder; speech-in-noise intelligibility
MeSH Terms: conditions — Auditory Perceptual Disorders | interventions — Hearing Aids

INTERVENTIONS:
Device: hearing aid, Phonak EduLink-FM System

SUMMARY:
In the management and remediation of students with specific performance deficits in speech-in-noise intelligibility, most often, a "triad" approach for treatment is used, which includes direct therapy, compensatory strategies, and environmental modifications.

The purpose of the study is to determine whether a new hearing aid, the Phonak EduLink-FM System, can improve specific performance deficits in speech-in-noise intelligibility. Participants will complete a test battery related to auditory processing, as well as some psychological tests and questionnaires. One group of participants with specific performance deficits in speech-in-noise intelligibility will receive the hearing aid for use in school; a second group will not. The effect of this treatment on auditory performance, school performance and satisfaction, attention and verbal learning and memory, self concept, behavior and listening effort following 26 weeks of hearing aid use will be compared across the groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of specific performance deficits in speech-in-noise intelligibility based on two or more standardized tests of auditory processing in noise including retests.
* Students in the 1st to 4th class of primary school

Exclusion Criteria:

* Hearing loss, defined as:

  * Air conduction pure tone thresholds (250-8000 Hz) exceeding 20 dBHL
  * Air-bone gaps, even in the presence of normal sensitivity, exceeding 10 dBHL
  * Abnormal tympanogram
* History or diagnosis of behavioral and/or emotional disorders meeting ICD-GM-criteria (including attention deficit/hyperactivity disorders (AD-/HD)
* Non-German speaking
* Cognitively impaired children (IQ < 85)
* Children currently using psychoactive medication
* Students with special education

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2005-03

PRIMARY OUTCOMES:
auditory performance | following 26 weeks hearing aid use
school performance and satisfaction | following 26 weeks hearing aid use
attention | following 26 weeks hearing aid use
verbal learning and memory | following 26 weeks hearing aid use

SECONDARY OUTCOMES:
self concept | following 26 weeks hearing aid use
behavior | following 26 weeks hearing aid use
listening effort | following 26 weeks hearing aid use

CONTACTS AND LOCATIONS:
Overall Officials: Peter Matulat, Principal Investigator — Department of Phoniatrics and Pediatric Audiology, University Hospital Münster; Antoinette G Dinnesen, Prof. Dr., Study Director — Department of Phoniatrics and Pediatric Audiology, University Hospital Münster
Locations (2):
- Department of Phoniatrics and Pediatric Audiology, University Hospital Münster, Münster, Germany
- Phonak AG, Stäfa, Switzerland